CLINICAL TRIAL: NCT01429831
Title: Aripiprazole for the Augmentation of Antidepressant Therapy: An Observational, Outpatients Study in Inadequate Responders Diagnosed With Major Depressive Disorder
Brief Title: Aripiprazole for the Augmentation of Antidepressant Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taiwan Otsuka Pharm. Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 031-TWB-1101i
Record Dates: First submitted 2011-09-01; First posted 2011-09-07 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Aripiprazole

ARMS (1):
- Aripiprazole (Experimental)
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — starting aripiprazole dose from 2-5mg/day, dose adjustment by every week, and maximum dose can up to 15mg/day. The duration is 6 weeks.

SUMMARY:
The study aims to evaluate effectiveness and tolerability of aripiprazole augmentation in outpatients with major depressive disorder who have had inadequate response to antidepressants in Taiwan clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients, either gender, 20-65 years of age
* Patients diagnosed with major depressive disorder as defined by Diagnostic and Statistical Manual of Mental Disorders (DSM-IV), who fulfill both the following criteria:

  * Having at least one and no more than three inadequate responses of antidepressants
  * HAM-D17 score ≥ 14
* Willing and able to comply with the study procedure and sign a written informed consent

Exclusion Criteria:

* Females who are pregnant/lactating or planning to be pregnant
* Presence of personality disorder cluster B (dramatic, emotional or erratic disorders) or any psychotic symptomatology in the current depressive episode based on Investigators judgment
* History of organic mental disorder within 1 year prior to the screening visit
* Acute risk of suicide attempts within 3 months prior to the initiation of study treatment (HAM D-17 score item 3 ≥ 3)
* Electroconvulsive therapy (ECT) for current episode
* Past exposure to aripiprazole treatment or any investigational product (including drug and invasive medical device) within 4 weeks prior to the initiation of study treatment
* History of substance / alcohol abuse within 1 year prior to the screening visit
* Patient with any medical or psychotic feature, including the presence of significant abnormal laboratory values, which is considered not suitable for this study by Investigator

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
17-Item Hamilton Depression Rating Scale (HAM-D17) score | Week 1, 2, 4 and 6
  Primary effectiveness endpoint:
  - Change from baseline in HAM-D17 score at Week 6
  Secondary effectiveness endpoints:
  1. Change from baseline in HAM-D17 score at Week 1, 2 and 4
  2. Response rate at Week 1, 2, 4 and 6
     - Response rate: decrease in HAM-D17 total score of at least 50%
  3. Remission rate at Week 1, 2, 4 and 6 - Remission rate: HAMD-17 score ≤ 7

SECONDARY OUTCOMES:
Clinical Global Impression of Severity (CGI-S) score | Week 1, 2, 4 and 6
  1. Change from baseline in CGI-S score at Week 1, 2, 4 and 6
  2. CGI-I score at Week 1, 2, 4 and 6
Sheehan Disability Scale (SDS) total score | Week 1, 2, 4 and 6
  Change from baseline in SDS total score at Week 1, 2, 4 and 6
World Health Organization Quality of Life (WHOQOL-BREF) score | Week 6
  Change from baseline in WHOQOL-BREF score at Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Te-Jen Lai, MD, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan